CLINICAL TRIAL: NCT00368342
Title: Chronic Bronchiolitis or Resistant Asthma?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baqiyatallah Medical Sciences University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S-340-14-6-1-PU-79
Record Dates: First submitted 2006-08-22; First posted 2006-08-24 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2006-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Erythromycin; Azithromycin; Clarithromycin

INTERVENTIONS:
Drug: Erythromycin, Azithromycin , Clarithromycin

SUMMARY:
Chronic Bronchiolitis or Resistant Asthma? Testing a way to diagnosis and treatment

ELIGIBILITY:
Inclusion Criteria:

* Difficult asthma

Exclusion Criteria:

* Patients with potential allergic bronchopulmonary aspergillosis i.e. with peripheral blood eosinophilia, sputum eosinophilia, or any sputum production and bronchiectasis
* A history of smoking
* Significant occupational or environmental exposures
* Evidence on emphysema on chest high resolution computed tomography (HRCT) scan

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Ghanei, Prof, Principal Investigator — Research Center of Chemical Injuries, Baqyatallah Medical Sciences University, Tehran, Iran